CLINICAL TRIAL: NCT04235530
Title: Comparison of Ultrasonography Guided Serratus Anterior Plane Block and Thoracic Paravertebral Block in Video-Assisted Thoracoscopic Surgery: A Prospective Randomized Double-blind Study
Brief Title: Comparison of Ultrasonography Guided Serratus Anterior Plane Block and Thoracic Paravertebral Block in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Merve Sena BAYTAR (Other Government)
Responsible Party: Sponsor-Investigator, Merve Sena BAYTAR, Medical Doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Other Study IDs: 2018-7/27
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
Keywords: thoracoscopic surgery video assisted; serratus anterior; paravertebral block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAS and DVAS: To measure the pain score of patients after surgery

SUMMARY:
The aim of this study is comparison of the effectiveness of ultrasound guided serratus anterior plane block and thoracic paravertebral block as a preventive analgesia method after VATS. Our secondary aim is to investigate patient and surgeon satisfaction, duration of block application, postoperative complications and hospital lenght of stay.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years
* ASA (American Society of Anesthesiologists) score I-II

Exclusion Criteria:

* inability to communicate
* body mass index (BMI) > 35 kg/m2
* infection in the area where the block was to be applied
* allergy to the drugs used
* mentally impaired
* bleeding impaired

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: who underwent elective video-assisted thoracoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
pain scores in rest and coughing | 24 hours
  Pain scores observed after surgery at 0, 1 ,2 ,6 ,12 ,24 th hours by visual analog scale. We assessed pain scores both in rest and coughing. This scale scores pain from 0 to 10. 0 means no pain and 10 means unbearable pain.
consumption of opioids | 24 hours
  We observed how much opioid ( how many miligrams) the patient consumed in 24 hours postoperatively with pca device.

SECONDARY OUTCOMES:
postoperative complications | 24 hours
  we compare postoperative complications like nausea, vomiting, constipation, pruritus first 24 hours after surgery.
lenght of hospital stay | 48 hours
  we compared how many days the patients stayed in the hospital until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Education and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No